CLINICAL TRIAL: NCT01583751
Title: Videoendoscopic Pilonidal Sinus Surgery. A New Technique
Brief Title: Videoendoscopic Pilonidal Sinus Surgery
Acronym: videosinus
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: SB Istanbul Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Erhan Aysan, Assoc Prof, SB Istanbul Education and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: pilonidal1
Record Dates: First submitted 2011-07-21; First posted 2012-04-24 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Recurrence; Postoperative Complication
Keywords: pilonidal sinus; new technique; videoendoscopic
MeSH Terms: conditions — Recurrence; Postoperative Complications; Pilonidal Sinus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- control (Experimental): excision and primer repair surgical technique will be perform
  Interventions: Procedure: videoendoscopic resection of pilonidal sinus

INTERVENTIONS:
Procedure: videoendoscopic resection of pilonidal sinus — Resection of pilonidal sinus tissue with videoendoscopic approach.
  Other Names: Active Comparator: Control: Group 1; Procedure/Surgery: Videoendoscopic: Group-2

SUMMARY:
This study examines performing pilonidal sinus surgery minimal invasively with videoendoscopic approach.

DETAILED DESCRIPTION:
Lots of surgical techniques are performing on pilonidal sinus disease treatment. Lately large flap techniques are popular but causing anatomical distortions and bad cosmesis. In this new approach the investigators concluded that two 1cm diameter holes are enough to surgical treatment. One hole is for videoendoscopic camera and the other one for grasper to extract piluses and granulation tissues.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic pilonidal sinus disease
* primer pilonidal sinus disease
* noncomplicated pilonidal sinus disease

Exclusion Criteria:

* Asymptomatic pilonidal sinus disease
* Recurrence pilonidal sinus disease
* complicated pilonidal sinus disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-03; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
recurrence rates | six months
  primary outcome measure of effectivity of pilonidal sinus surgery is recurrence rates.

SECONDARY OUTCOMES:
postoperative complications, wound healing | 1 month
  Postoperative complications such as bleeding and infection are important outcome measurements. Wound healing time is the other important one.

CONTACTS AND LOCATIONS:
Overall Officials: erhan aysan, assoc prof, Study Director — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)